CLINICAL TRIAL: NCT06651242
Title: Effectiveness Evaluation on the Decision Preferences and Decision Support Intervention of Minor Cancer Patients and Their Parents
Brief Title: Decision Support Intervention of Minor Cancer Patients and Their Parents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KMUHIRB- SV(II)-20220022
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Pediatric Cancer; Adolescent Health; Decision Aids; Parents of Children With Cancer; Decision Making ,Shared
Keywords: Minor Cancer; Parents; Decision Preferences; Decision Support; Intervention
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Decision-making information aids (Experimental)
  Interventions: Other: Decision-making information aids
- Routine care (Sham Comparator)
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Decision-making information aids — Provide a decision-making information aids to assist patients and their parents in treatment decision making.
  Arms: Decision-making information aids
Other: Routine care — Routine care
  Arms: Routine care

SUMMARY:
The purpose of this stuidy are: (1) to explore the information needs of parents having children with cancer when making treatment decisions; (2) to develop a Taiwan version of the Control Preferences Scale for decision support aids; (3) to implement and evaluate the effectiveness of involving minor cancer patients and their parents in treatment decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for Parents:

  1. Age over 20 years.
  2. Child under 20 years old, diagnosed with cancer by a doctor.
  3. their child know her/his cancer diagnosis.
  4. Agree to have the child participate in family meeting and have ability to communicate in Mandarin or Taiwanese.
* Inclusion Criteria for Minors:

  1. Aged between 7 and 20 years, diagnosed with pediatrtic cancer.
  2. Aware of their cancer diagnosis.
  3. Able to express their thoughts to the researcher in Mandarin or Taiwanese.
  4. Both the minor and their legal guardian consent to participate in the study.

Exclusion Criteria:

1. Diagnosed with depression, and/or anxiety, and/or other mental disorders.
2. Legal guardian is unwilling to inform the minor of their diagnosis.
3. Minor is unwilling to share their thoughts with their parents.

Ages: 7 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Exploring decision-making preferences among parents and minor using the Control Preferences Scale (CPS) | baseline and 1.3.6 months
  The CPS is a method for assessing individual preferences in medical decision-making roles, consisting of five options that represent five different roles. (A) I prefer to make the decision about which treatment I will receive, (B) I prefer to make the final decision about my treatment after seriously considering my doctor's opinion, (C) I prefer that my doctor and I share responsibility for deciding which treatment is best for me, (D) I prefer that my doctor makes the final decision about which treatment will be used, but seriously considers my opinion, (E) I prefer to leave all decisions regarding treatment to my doctor. The five responses are classified into three categories representing active(A and B), collaborative (C) and passive (D and E) decision-making preference.
Exploring the perceived involvement in decision-making among parents and minor using the Perceived Involvement in Care Scale (PICS) | baseline and 1.3.6 months
  This scale comprises 13 items and is divided into three subscales, which measure physician facilitation (4 items), patient information acquisition (4 items), and patient decision-making involvement (4 items). A 5-point Likert scale is used, where higher scores indicate greater perceived involvement in decision-making.
Exploring decision-making experiences of parents and minor using the Decision Conflict Scale (DCS) | baseline and 1.3.6 months
  This scale consists of 16 items, with the first 12 items assessing decision experiences, including uncertainty, understanding of information, unclear values, support during the decision-making process, and satisfaction with decisions. It uses a 5-point Likert scale, with higher scores indicating greater decision conflict.
Exploring perceived family adaptability and cohesion among parents and minor using the Family Adaptability and Cohesion Evaluation Scales IV (FACES IV) | baseline and 1.3.6 months
  The evaluation of family functioning involves: (1) Balanced Scales: Cohesion and Flexibility, (2) Unbalanced Scales: Disengaged, Enmeshed, Rigid, and Chaotic, (3) Family Communication, and (4) Family Satisfaction. The instrument consists of eight subscales with a total of 62 items, rated on a five-point Likert scale. The Family Cohesion and Flexibility scales include 42 items (0-42), divided into six sections with scores ranging from 7 to 35 per section. The Family Communication scale, which assesses positive communication and openness, contains 10 items (43-52) with scores ranging from 10 to 50. The Family Satisfaction scale, measuring satisfaction with cohesion, flexibility, and communication, also has 10 items (53-62), scoring from 10 to 50. Higher scores on Cohesion and Flexibility suggest a healthier family system; higher scores on Disengaged, Enmeshed, Rigid, and Chaotic indicate dysfunction; higher scores on Communication and Satisfaction denote more positive perceptions.
Exploring minor' coping behaviors in response to illness and treatment using the Paediatric Cancer Coping Scale | baseline and 1.3.6 months
  This scale consists of 33 items, scored from 0 ("never") to 3 ("often"). Higher scores indicate more frequent coping behaviors.
Exploring minor' anxiety levels using the Revised Children's Manifest Anxiety Scale-2 (RCMAS-2) | baseline and 1.3.6 months
  This 49-item scale assesses four dimensions: defensiveness, physiological anxiety, worry, social anxiety, and performance anxiety. Responses are either "yes" (indicating the presence of a symptom) or "no" (indicating the absence of a symptom).
Exploring parental anxiety under different characteristics using the State-trait anxiety inventory (STAT) | baseline and 1.3.6 months
  This scale consists of 20 items measuring individual anxiety traits under different characteristics. It uses a 4-point Likert scale, with higher scores indicating higher levels of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No